CLINICAL TRIAL: NCT04979026
Title: Clinical Investigation of a Novel Approach for the Prevention of Deep Venous Thrombosis After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ming-Chou Ku, Principal Investigator, Show Chwan Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RB19013
Record Dates: First submitted 2021-07-06; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Deep Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active ankle pumping without any reminders (No Intervention): In group 1, active ankle pumping exercise for the operative limb was performed without any reminder during hospitalization and at home after being discharged.
- intermittent pneumatic compression (Active Comparator): In group 2, intermittent pneumatic compression was applied to the operative low limb during hospitalization, while active ankle pumping exercise was adopted without any reminder after discharge.
  Interventions: Device: intermittent pneumatic compression
- active ankle pumping with a regular watch alarm (Experimental): In group 3, in addition to the active ankle pumping exercise for the operative limb, the patients were reminded to exercise at specific time points with a vocal alarm and vibration through a wrist watch during the hospitalization period and at home after discharge. The watch was continuously used until the 14th day when the patients returned to the hospital for examination.
  Interventions: Device: active ankle pumping with a regular watch alarm

INTERVENTIONS:
Device: active ankle pumping with a regular watch alarm — In addition to the active ankle pumping exercise for the operative limb, the patients were reminded to exercise at specific time points with a vocal alarm and vibration through a wrist watch during the hospitalization period and at home after discharge.
  Arms: active ankle pumping with a regular watch alarm
Device: intermittent pneumatic compression — In this group, intermittent pneumatic compression was applied to the operative low limb during hospitalization, while active ankle pumping exercise was adopted without any reminder after discharge.
  Arms: intermittent pneumatic compression

SUMMARY:
Venous thromboembolism, including deep vein thrombosis (DVT), has long been recognized as the most frequent complication within 7 to 14 days after orthopedic surgery, especially total joint arthroplasty. Without prophylactic therapy, the incidence of DVT and pulmonary embolism reaches up to 60% following orthopedic surgery. The possible damage to the vessel wall during the operation, the venous stasis caused by long-term bed rest, and the hypercoagulability of the blood after the surgery are the 3 main reasons for the formation of DVT. In most cases, the thrombi resolve spontaneously; however, some of them (about 1~4%) may develop into symptomatic and even fatal DVT.

Ankle pumping exercise is currently suggested for the patients with joint placement surgery to prevent the formation of lower-extremity DVT after orthopedic surgery. However, the compliance of the exercise at home is unclear. In order to remind the patients to the active ankle exercise and record the executive rate, a device was developed to help the patient to exercise in the hospital and at home. The device will remind the patient to exercise at specific time point by verbal and vibrations, and detect the range of motion during the exercise for further analysis. The aim of this study is to access the effect of a non-invasive novel device in preventing the formation of lower limb DVT. Maximum venous outflow, maximum venous capacity, and blood rheology were measured and the incidence of DVT was recorded for the data analysis.

DETAILED DESCRIPTION:
Background. Deep vein thrombosis (DVT) has long been recognized as the most frequent complication that occurs 7-14 days after total knee replacement (TKR). Physical therapy, including active ankle pumping exercises and intermittent pneumatic compression, is suggested for the prevention of DVT. However, the exercise implementation rate is not clear, particularly at home. In order to remind the patients to exercise after TKR, a watch with voice and vibration alarms at the set time was used.

Objective The first aim of this study was to compare the effect of active ankle movement with and without reminders on the prevention of DVT. The second aim was to compare the difference in the effect of intermittent pneumatic compression and active ankle movement on the prevention of DVT.

Design. A Pilot Randomized Controlled Trial Methods. The patients were divided into three groups according to the therapeutic protocols. The patients in group 1 conducted active ankle pumping without any reminders, those in group 2 underwent intermittent pneumatic compression, and those in group 3 conducted active ankle pumping with a regular watch alarm. The parameters of blood flow, namely peak flow velocity and flow volume, in the bilateral common femoral vein and popliteal vein on the 1st, 3rd, and 14th days after surgery were measured using the echo technique, as an index to evaluate the effect of DVT prevention among the three groups.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent total knee replacement surgery

Exclusion Criteria:

* Patients with a history of cardiovascular disease, such as DVT, dyslipidemia, hypertension, myocardial infarction, and hemorrhagic disease were excluded from this study.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
change of peak flow velocity | The peak flow velocity was determined on the 1st, 3rd, and 14th days after surgery.
  The peak flow velocity was directly detected using the Doppler images. The examination was conducted by an experienced technician.
change of flow volume | The flow volume was determined on the 1st, 3rd, and 14th days after surgery.
  The flow volume was directly detected using the Doppler images. The examination was conducted by an experienced technician.
Number of Participants with stasis | Stasis was determined on the 1st, 3rd, and 14th days after surgery.
  Venous stasis was determined by a peak flow velocity lower than 10 cm/s, and the color of the blood inside the vein represented in the echo image was gray. In addition, the contour of the vein was compressible under a slight compression force with an echo transducer.
Number of Participants with deep venous thrombosis | Deep venous thrombosis was determined on the 1st, 3rd, and 14th days after surgery.
  If the peak blood flow, flow volume, and blood echo image were the same as that of stasis, but the contour of the vein was incompressible under a slight compression, the cases were recorded as deep venous thrombosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson DR, Dunbar M, Murnaghan J, Kahn SR, Gross P, Forsythe M, Pelet S, Fisher W, Belzile E, Dolan S, Crowther M, Bohm E, MacDonald SJ, Gofton W, Kim P, Zukor D, Pleasance S, Andreou P, Doucette S, Theriault C, Abianui A, Carrier M, Kovacs MJ, Rodger MA, Coyle D, Wells PS, Vendittoli PA. Aspirin or Rivaroxaban for VTE Prophylaxis after Hip or Knee Arthroplasty. N Engl J Med. 2018 Feb 22;378(8):699-707. doi: 10.1056/NEJMoa1712746. PMID 29466159
- [Background] Blagojevic M, Jinks C, Jeffery A, Jordan KP. Risk factors for onset of osteoarthritis of the knee in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2010 Jan;18(1):24-33. doi: 10.1016/j.joca.2009.08.010. Epub 2009 Sep 2. PMID 19751691
- [Background] Boylan MR, Perfetti DC, Kapadia BH, Delanois RE, Paulino CB, Mont MA. Venous Thromboembolic Disease in Revision vs Primary Total Knee Arthroplasty. J Arthroplasty. 2017 Jun;32(6):1996-1999. doi: 10.1016/j.arth.2016.12.051. Epub 2017 Jan 11. PMID 28209273
- [Background] Changulani M, Kalairajah Y, Peel T, Field RE. The relationship between obesity and the age at which hip and knee replacement is undertaken. J Bone Joint Surg Br. 2008 Mar;90(3):360-3. doi: 10.1302/0301-620X.90B3.19782. PMID 18310761
- [Background] Chen Q, Huang S, Chen X, Feng L, Zhu X. [Clinical efficacy of multi-pattern detumescence after total knee arthroplasty treated with acupoint massage and mild moxibustion]. Zhongguo Zhen Jiu. 2016 May;36(5):471-5. Chinese. PMID 27509603